CLINICAL TRIAL: NCT00495924
Title: Prognostic Relevance of Perioperative Cancer Cell Dissemination and Systemic Immune Suppression in Resectable Ductal Pancreatic Adenocarcinoma
Brief Title: Perioperative Cancer Cell Dissemination and Systemic Immune Suppression in Resectable Ductal Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Topal Baki, MD, PhD, Katholieke Universiteit Leuven
Other Study IDs: 3M070038; G.0635.07
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Pancreatic Neoplasms; Adenocarcinoma; Neoplasm Circulating Cells; Tumor Markers, Biological; Monitoring, Immunologic
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, serum, blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PD: Patients undergoing pancreaticoduodenectomy for pancreatic or peri-ampullary tumours.
  Interventions: Procedure: Pancreatic resection (PD)

INTERVENTIONS:
Procedure: Pancreatic resection (PD) — PD is a standard therapeutic surgical procedure. No additional interventions are performed.

SUMMARY:
The purpose of this study is to determine whether early recurrence after curative resection of ductal pancreatic adenocarcinoma can be explained by either dissemination of cancer cells during intraoperative tumour manipulation, post-operative systemic immune suppression, alteration of biological properties of circulating cancer cells or a combination of these.

DETAILED DESCRIPTION:
Prognostic relevance of circulating cancer cells and immunosuppression in resectable pancreatic carcinoma

1. Introduction

   Pancreatic adenocarcinoma is the fourth commonest cause of death from cancer in men and women, with 5-year survival for all stages of disease of less than 5%. The case-fatality rate for pancreatic cancer is extremely high and virtually identical to the number of new cases (World Health Organization. World cancer report. Lyon: IACR Press; 2003). Most patients with cancer of the pancreas are diagnosed at an advanced stage and have a median survival of 4 to 10 months, depending on the extent of disease and irrespective the type of treatment modality. Overall, fewer than 5% of the patients have resection with curative intent, though over 80% will develop cancer recurrence (Jemal A, Thomas A, Murray T, Thun M. Cancer Statistics. CA Cancer J Clin 2002; 52: 23-47). The primary site of metastatic disease in patients with pancreatic cancer is the liver and/or the peritoneal cavity.

   Cancer recurrence is multifactorial and determined by patient-, tumour-, and surgery-related factors. Any combination of several mechanisms have been proposed by which cancer may recur following potentially curative resection (Coffey JC, Wang JH, Smith MJF, Bouchier-Hayes D, Cotter TG,and Redmond HP. Excisional surgery for cancer cure: therapy at a cost. Lancet Oncol 2003;4:760-68). Surgery may contribute to the overall residual tumor burden by adding disseminated cancer cells during tumor manipulation. Due to post-operative immunosuppression the patient may become more susceptible to tumorigenesis and/or disseminated cancer cells may escape the immune response more easily. Finally, surgical resection may alter biological properties of cancer cells and lead to increased cellular proliferation and reduced cell death.
2. Cancer cell dissemination

   Solid markers are lacking to predict cancer recurrence or cancer progression before being measurable with conventional or modern diagnostic imaging. Molecular techniques such as the reverse transcriptase polymerase chain reaction (RT-PCR) technique have proven to be a highly sensitive method and a powerful tool in the study of cancer metastasis (Raj GV, Moreno JG, Gomella LG. Utilization of Polymerase Chain Reaction Technology in the Detection of Solid Tumors. Cancer 1998; 82: 1419-42). The prognostic relevance of circulating cancer cells in patients with pancreatic cancer is hardly studied. In patients with breast cancer the number of circulating cancer cells expressing EpCAM (epithelial cell adhesion molecule) has proven to be an independent predictor of progression-free and overall survival (Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med 2004; 351: 781-91). EpCAM is a marker present on most epithelial cell tumours and frequently overexpressed in primary and metastatic adenocarcinoma including pancreatic cancer (Rao CG, Chianese D, Doyle GV, Miller MC, Russell T, Sanders RA Jr, Terstappen LW. Expression of epithelial cell adhesion molecule in carcinoma cells present in blood and primary and metastatic tumors. Int J Oncol 2005; 27: 49-57). Also, other markers such as CEA, CK20, K-ras have been used to detect disseminated pancreatic cancer cells. In patients with colorectal carcinoma circulating cancer cells in peripheral or in mesenteric venous blood as detected by RT-PCR, using CEA and CK20 mRNA transcripts, seem to represent a prognostic factor (Yamaguchi K, Takagi Y, Aoki S, Futamura M, Saji S. Significant detection of circulating cancer cells in the blood by reverse transcriptase-polymerase chain reaction during colorectal cancer resection. Ann Surg 2000; 232: 58-65. Guller U, Zajac P, Schnider A, Bösch B, Vorburger S, Zuber M, Spagnoli GC, Oertli D, Maurer R, Metzger U, Harder F, Heberer M, Marti WR. Disseminated single tumor cells as detected by real-time quantitative polymerase chain reaction represent a prognostic factor in patients undergoing surgery for colorectal cancer. Ann Surg 2002; 236: 768-76).
3. Molecular characteristics of metastatic cancer cells

   The development of metastasis is a highly selective process favoring the survival of a minor subpopulation of metastatic cells. To produce metastases, tumor cells from this subpopulation must complete a sequence of interrelated steps. To produce clinically relevant distant metastases, the successful metastatic cell must therefore exhibit a complex phenotype that is regulated by transient or permanent changes at the gene level. Many malignant tumors, including pancreatic cancer, contain heterogeneous subpopulations of cells. This heterogeneity is exhibited in a wide range of genetic, biochemical, immunological, and biological characteristics such as growth rate, antigenic and immunogenic status, cell surface receptors and products, enzymes, karyotypes, cell morphologies, invasiveness, drug resistance, and metastatic potential. It is likely that specific tumor cells or colonies within the larger heterogeneous tumor specimen are the forerunners of distant metastases. The overall efficiency of the whole metastatic process itself is low. Although the absolute number of cancer cells required for metastasis in humans is unknown, a positive relationship between the number of circulating cancer cells and the subsequent development of metastases has been the subject of several experimental studies (Fisher, E.R. and Fisher, B. Experimental study of factors influencing development of hepatic metastases from circulating tumor cells. Acta Cytol. 9: 146-159, 1965. Fidler, I.J. The relationship of embolic homogeneity, number, size and viability to the incidence of experimental metastasis. Europ. J. Cancer 9: 223-227, 1973. Liotta, L.A., Kleinerman, J., Saidel, G. Quantitative relationships of intravascular tumor cells, tumor vessels and pulmonary metastasis. Cancer Res. 34: 977-1004, 1974. Weiss, L., Mayhew, E., Glaves, R.P. and Holmes, J.C. Metastatic inefficiency in mice bearing B16 melanomas. Br. J. Cancer 45: 44-53, 1982. Topal B, Aerts JL, Roskams T, Fieuws S, Van Pelt J, Vandekerckhove P, Penninckx F. Cancer cell dissemination during curative surgery for colorectal liver metastases. Eur J Surg Oncol 2005; 31: 506-511).

   The poor prognosis and lack of effective treatments for pancreatic cancer arise from several causes. There are currently no effective biomarkers useful for early detection of pancreatic cancer that tends to rapidly invade surrounding structures and undergo early metastatic spreading. Moreover, pancreatic cancer is highly resistant to both chemotherapy and radiation therapy. Currently, the molecular basis for these characteristics is unknown. Gene expression profiles provide important information about the molecular characteristics of the cancers and can be used to distinguish closely related cancer subtypes. Gene profiling can also be used to develop candidate biomarkers and to identify groups of genes involved in specific functional aspects of tumor biology. Gene expression profiles that could distinguish between pancreatic tumors, chronic pancreatitis and normal pancreatic tissue have been studied extensively using different microarrays and microarray platforms. The differentially expressed genes in pancreatic tumor tissues were found to be quite specific and highly reproducible among platforms and studies (Crnogorac-Jurcevic T, Efthimiou E, Nielsen T, Loader J, Terris B, Stamp G, Baron A, Scarpa A and Lemoine NR. Expression profiling of microdissected pancreatic adenocarcinomas. Oncogene 2002; 21: 4587-4594. Han H, Bearss DJ, Browne LW, Calaluce R, Naagle RB, Von Hoff DD. Identification of differentially expressed genes in pancreatic cancer cells using cDNA microarray. Cancer Res 2002; 62: 2890-96. Iacobuzio-Donahue CA, Ashfaq R, Maitra A, Adsay NV, Shen-Ong GL, Berg K, Hollingsworth MA, Cameron JL, Yeo CJ, Kern SE, Goggins M, Hruban RH. Cancer Res 2003; 63: 8614-22. Logsdon CD, Simeone DM, Binkley C, Arumugam T, Greenson JK, Giordano TJ, Misek DE, Hanash S. Molecular profiling of pancreatic adenocarcinoma and chronic pancreatitis identifies multiple genes differentially regulated in pancreatic cancer. Cancer Res 2003; 63: 2649-57).
4. Peri-operative immunological changes

   Suppression of the immune system is a feature of the post-operative stress response, in which natural killer (NK) and lymphocyte activated killer (LAK) cells form an integral component in immune anti-tumor surveillance. However, a tumor type-specific immune reaction in pancreatic cancer or in patients undergoing surgery is lacking. Anti-tumoral activities of NK and LAK cells are reduced immediately after surgery so the additive effects of surgery may be sufficient to improve the ability of disseminated cancer cells to evade the host immune response long enough for metastases to develop (Da Costa ML, Finnegan N, Flynn M, Bouchier-Hayes DJ. Laparotomy and laparoscopy differentially accelerate experimental flank tumourgrowth. Br J Surg 1998; 85: 1439-42.) (Da Costa ML, Redmond HP, Bouchier-Hayes DJ. The effect of laparotomy and laparoscopy on the establishment of spontaneous tumour metastases. Surgery 1998; 124: 516-26).

   The suppressive immunological changes that follow surgical stress occur along a temporal pattern. Depression of cellular immunity to tumor-associated antigen and depression of delayed-type hypersensitivity are present for up to 3 weeks after surgery. In patients with pancreatic cancer the prevalence of regulatory T cells (Treg) is increased in the peripheral blood as well as in the tumour microenvironment. These Treg cells (CD4+25+) are phenotypically similar to Treg cells from normal donors by coexpression of CD45R0 and CTLA-4 molecules as well as cytokine profile. Regulatory CD4+25+ lymphocytes infiltrate tumor and regional lymph nodes, and suppress activation of CD8+ lymphocytes and helper CD4+25- lymphocytes (Liyanage, U. K., T. T. Moore, H. G. Joo, Y. Tanaka, V. Herrmann, G. Doherty, J. A. Drebin, S. M. Strasberg, T. J. Eberlein, P. S. Goedegebuure, and D. C. Linehan. 2002. Prevalence of regulatory T cells is increased in peripheral blood and tumor microenvironment of patients with pancreas or breast adenocarcinoma. J Immunol 169:2756).

   However, the oncological significance of changes in activities and numbers of NK, LAK, Treg and dendritic cells still has to be confirmed.
5. Aims / Endpoints

   * Is the number of circulating cancer cells a determinant for cancer recurrence and/or survival following potentially curative resection of pancreatic cancer?
   * Is the genetic profile of circulating cancer cells a determinant for cancer recurrence and/or survival following potentially curative resection of pancreatic cancer?
   * Is peri-operative immunosuppression correlated with cancer recurrence and/or survival following potentially curative resection of pancreatic cancer?
6. Patient selection and inclusion criteria: Potentially curable/ resectable pancreatic cancer
7. Study interventions

   - Quantitative analysis of circulating cancer cells

   In the present study peripheral venous blood samples will be obtained before the start of surgery, at the end of surgery, on the first day after and on day 7 after surgery through a central venous catheter. Tumour tissue samples and random liver tru-cut biopsies will be obtained intra-operatively. Real-time quantitative RT-PCR technique (TaqManR), based on 3 different target markers (CEA, CK20 and EpCAM mRNA transcripts) and beta-glucuronidase (GUS) as control gene, will be used to detect and quantify circulating cancer cells in the blood stream. Normalized copy numbers (NCN) will be determined in each sample (analyzed in duplicate). RNA extraction from all samples will be performed using RNeasy mini kit(Qiagen, BD Company). Sample preparation, cDNA synthesis and PCR will be performed in separated rooms in order to prevent cross-contamination.

   - Genetic profiling of disseminated cancer cells

   Oligonucleotide microarray analysis of mRNA extracted from the primary pancreatic tumor and from disseminated cancer cells before, during and the day after surgery. The focus of this study is not to identify specific markers for diagnosis or for drug targets but to find indications of metastasis through the study of gene expression in cancer cells circulating in the bloodstream. Our main objective is to analyze expression profiles of circulating pancreatic cancer cells. Changes will be analyzed in the expression of genes representative of several different pathways frequently altered during the progression of cancer such as tumor suppressors, oncogenes, signal transduction molecules, growth factors and angiogenesis factors. Gene expression profile data will be obtained on apoptosis, cell cycle, cell growth and differentiation, cell migration and motility, signal transduction and other cancer-related genes. Latest developments in microarray technology comprise the manufacturing of the complete genome and in designing new amplification strategies to be able to analyze very small samples less than 1 ng total RNA (Xiang CC, Chen M, Kozhich OA, Phan QN, Inman JM, Chen Y, Brownstein MJ. Probe generation directly from small number of cells for DNA microarray studies. Biotechniques 2003; 34: 386-8, 390, 392-3. Schindler H, Wiese A, Auer J, Burtscher H. cRNA target preparation for microarrays: comparison of gene expression profiles generated with different amplification procedures. Anal Biochem 2005; 344: 92-101. Puskás LG, Zvara Á, Hackler L Jr, Van Hummelen P. RNA amplification results in reproducible microarray data with slight ratio bias. Biotechniques 2002; 32: 1330-1341). In the present study the number of cancer cells circulating in the blood stream is expected to be extremely small. Therefore, linear RNA amplification (T7 RNA-polymerase) is used in order to generate enough material for labeling and hybridization on the arrays. Two rounds of amplification are performed routinely. This has been performed successfully and reproducibly starting from as little as 700 cells isolated via Laser Capture Microdissection (data unpublished).

   - Preparation of cell suspension microarrays to isolate circulating cancer cells.

   Although most of the microarray challenges are known and under control, the present study has an important specific challenge that is the isolation and enrichment of the circulating cancer cells. Currently, the proportion of circulating cancer cells to other nucleated blood cells (leucocytes) is unknown in patients suffering from pancreatic cancer. Therefore, the first step will be to determine the number of cancer cells per ml blood in pancreatic cancer patients and to determine the variability among different patients. A second step is to develop an enrichment method to concentrate the cancer cells without selecting specific types of cancer cells or loss of information on the initial proportion of cancer cells in each patient's blood stream. The fastest way to isolate the circulating cancer cells is using flow cytometry after density-gradient pre-enrichment in combination with negative selection strategies to discard leukocytes (CD45+ and CD34+) from the sorted 'circulating' cancer cells. Isolating cells with LCM has been used many times successfully for microarray studies. It has been reported that LCM can easily dissect several thousands of cells from pancreatic tissue with a RNA-yield of around 1ng/1000 cells (Datson NA, Meijer L, Steenbergen PJ. Morsiak MC, van der Laan S, Meijer OC, de Kloet ER. Expression profiling in laser-microdissected hippocampal subregions in rat brain reveals large subregion specific differences in expression. Eur J Neurosci 2004; 20: 2541-54. Player A, Barrett JC, Kawasaki ES. Laser capture microdissection, microarrays and the precise definition of a cancer cell. Expert Rev Mol Diagn 2004; 4: 831-40. Espina V, Geho D, Mehta AI, Petricoin EF 3rd, Liotta LA, Rosenblatt KP. Pathology of the future: molecular profiling for targeted therapy. Cancer Invest 2005; 23: 36-46. Crnogorac-Jurcevic T, Efthimiou E, Nielsen T, Loader J, Terris B, Stamp G, Baron A, Scarpa A and Lemoine NR. Expression profiling of microdissected pancreatic adenocarcinomas. Oncogene 2002; 21: 4587-4594).

   - Immunological changes

   Since a tumor type-specific immune reaction in pancreatic cancer or in patients undergoing surgery is lacking, the present study will assess the systemic immunological changes including cytokine levels before and at different time intervals following potentially curative surgery in pancreatic cancer patients.

   PBMC will be extracted from peripheral venous blood and used for further analysis under FACS (fluorescence-activated cell sorter) to determine the prevalence of:
   * CD3-19+ (B-lymphocytes)
   * CD3+56+ (Killer cells)
   * CD3-56+CD16+ (NK natural killer cells)
   * CD8+ (Cytotoxic T-lymphocytes)
   * CD4+25- (Helper T-lymphocytes)
   * CD4+25+127- (Regulatory T-lymphocytes)
   * Inflammatory cytokines in peripheral blood (IL-1b, IL-6, IL-8, IL-10, IL-12 and TNF) will be analysed using a commercially available 'BD Cytometric Bead Array (CBA) Human Inflammatory Kit'.
   * PBMC (peripheral blood mononuclear cells) and tumour tissue will be stored in liquid nitrogen for analysis in future studies.
8. Statistical analysis

   Univariate analysis as well as corrected, multivariate analysis will be performed in order to identify the optimally combined prognostic group of factors: patient-, tumour-, and treatment-associated factors as well as the amounts of disseminated cancer cells, their genetic expression profile and immunological changes following surgery. The events to study will be cancer recurrence (disease free survival DFS) and death (overall survival OS).
9. Expected patient accrual "Single center study": UZ.Gasthuisberg - KU.Leuven, Belgium Expected annual patient registration: 30 pts / year Duration of patient accrual: 2 years

ELIGIBILITY:
Inclusion Criteria:

* Suspected ductal pancreatic adenocarcinoma (pathological confirmation required after resection of tumour);
* Informed consent.

Exclusion Criteria:

* Any malignant tumour within 5 years prior to pancreatic resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pancreaticoduodenectomy for pancreatic or peri-ampullary tumours.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, PhD, Study Director — Catholic University Leuven, Belgium; Gregory Sergeant, MD, Principal Investigator — Catholic University Leuven
Locations (1):
- Department of Abdominal Surgery, Catholic University Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Sergeant G, van Eijsden R, Roskams T, Van Duppen V, Topal B. Pancreatic cancer circulating tumour cells express a cell motility gene signature that predicts survival after surgery. BMC Cancer. 2012 Nov 16;12:527. doi: 10.1186/1471-2407-12-527. PMID 23157946
- [Derived] Sergeant G, Roskams T, van Pelt J, Houtmeyers F, Aerts R, Topal B. Perioperative cancer cell dissemination detected with a real-time RT-PCR assay for EpCAM is not associated with worse prognosis in pancreatic ductal adenocarcinoma. BMC Cancer. 2011 Jan 31;11:47. doi: 10.1186/1471-2407-11-47. PMID 21281486